CLINICAL TRIAL: NCT04458324
Title: Hybrid Functional Electrical Stimulation Exercise to Prevent Cardiopulmonary Declines in High-level Spinal Cord Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, Director, Cardiovascular Research Lab, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2020P001363
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries
Keywords: Function Electrical Stimulation (FES)-Rowing
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Buspirone; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to one of four groups with equal chance: 1. NIV + Buspar, 2. NIV + placebo, 3. sham NIV + Buspar, or 4. sham NIV + placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- NIV + Buspar (Experimental): Subjects will perform 6 months of FES-row-training while receiving NIV and taking Buspar.
  Interventions: Drug: Buspirone Hydrochloride; Device: Noninvasive Ventilation (NIV); Other: Functional Electrical Stimulation Row Training (FESRT)
- NIV + placebo (Placebo Comparator): Subjects will perform 6 months of FES-row-training while receiving NIV and taking placebo.
  Interventions: Drug: Buspirone placebo; Device: Noninvasive Ventilation (NIV); Other: Functional Electrical Stimulation Row Training (FESRT)
- sham NIV + Buspar (Sham Comparator): Subjects will perform 6 months of FES-row-training while receiving sham NIV and taking Buspar.
  Interventions: Drug: Buspirone Hydrochloride; Device: Sham Non-invasive ventilation (NIV); Other: Functional Electrical Stimulation Row Training (FESRT)
- sham NIV + placebo (Active Comparator): Subjects will perform 6 months of FES-row-training while receiving sham NIV and taking placebo.
  Interventions: Drug: Buspirone placebo; Device: Sham Non-invasive ventilation (NIV); Other: Functional Electrical Stimulation Row Training (FESRT)

INTERVENTIONS:
Drug: Buspirone Hydrochloride — Subjects take 30 mg buspirone HCl twice a day for 6 months.
  Other Names: Buspar
  Arms: NIV + Buspar; sham NIV + Buspar
Drug: Buspirone placebo — Subjects take a placebo tablet twice a day for 6 months.
  Arms: NIV + placebo; sham NIV + placebo
Device: Noninvasive Ventilation (NIV) — The ventilator will be set in spontaneous mode with a ramp to reach a minimal pressure of 12 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Arms: NIV + Buspar; NIV + placebo
Device: Sham Non-invasive ventilation (NIV) — The ventilator will be set in spontaneous mode with a ramp to reach a maximal pressure of 5 centimeters of water (cmH2O) during inspiration and 3 cmH2O during expiration.
  Arms: sham NIV + Buspar; sham NIV + placebo
Other: Functional Electrical Stimulation Row Training (FESRT) — Subjects participate in a supervised exercise training program 2-3 times/week for 6 months using an adapted indoor rower and FES.

SUMMARY:
Over the past ten years, the Cardiovascular Research Laboratory at Spaulding has refined a unique form of exercise for those with spinal cord injuries (SCI). Functional Electrical Stimulation Row Training (FESRT) couples volitional arm and electrically controlled leg exercise, resulting in the benefits of large muscle mass exercise. However, despite the potential for enhancing aerobic capacity by training the denervated leg skeletal muscle via hybrid FES exercise, the inability to increase ventilation beyond limits set by high level SCI restricts aerobic capacity.

This research study will investigate two potential methods of improving ventilation in those with high-level SCI through a double-blind randomized trial. One method is non-invasive ventilation (NIV), which is an external breathing support machine. The second method is the use of Buspar, a drug, which has been used to treat respiratory dysfunction after SCI in rats and some human case reports.

In this study, participants will engage in a 6-month FES row training program while receiving either NIV or shamNIV and Buspar or placebo, and under study tests to evaluate cardiopulmonary health and fitness.

DETAILED DESCRIPTION:
Regular aerobic exercise with sufficient intensity can improve overall health, however daily energy expenditure is low in those with SCI, especially in those with high level lesions. The investigators have developed Functional Electrical Stimulation Row Training (FESRT) that couples volitional arm and electrically controlled leg exercise, increasing the active muscle and resulting in benefits of large muscle mass exercise. Despite the potential for enhancing aerobic capacity, those with high level lesions (T3 and above) have a remaining obstacle to attaining higher work capacities: a level of pulmonary muscle denervation. The investigators preliminary work suggests this limits the aerobic capacity that can be achieved with FESRT.

External ventilatory support could improve the ability to exercise train and hence enhance the adaptations to chronic exercise in high level SCI. Non invasive ventilation (NIV) during exercise training has been shown to improve gains in exercise capacity in those with similarly restrictive breathing. Therefore, the investigators hypothesize that the use of NIV during FESRT will reduce ventilatory limits to exercise, leading to increased aerobic capacity in high level SCI. In addition, pharmacologic treatments may augment respiratory control and improve exercise ventilatory responses. Buspirone can reverse respiratory abnormalities consequent to SCI in rats, and humans case reports suggest successful Buspirone treatment of respiratory dysfunction

Therefore, the investigators propose a double-blind 2x2 trial of 6 months of FESRT with NIV or Sham and Buspirone or Placebo in individuals with acute, high-level SCI. The investigators hypothesize that both NIV and Buspirone will improve ventilatory exercise responses and that combined treatment will have the greatest effect. This will result in greater improvements in aerobic capacity and concomitant increases in pulmonary function and reductions in cardiometabolic risk. This work proposes two approaches to overcome ventilatory limitations to exercise in high level SCI and allow for greater improvements in cardiopulmonary capacity - one that overcomes mechanical limitations of paralyzed pulmonary musculature and one that treats loss of serotonergic respiratory control, both of which may contribute to blunted ventilatory responses. The ultimate purpose of this research is to optimize exercise for a population that both needs and seeks the broad range of benefits that exercise can confer.

ELIGIBILITY:
Inclusion Criteria:

* SCI outpatients aged 18-45 years
* medically stable
* body mass index 18.5-30 kg/m2 to include normal to overweight but not obese individuals
* 3-months to 6-years post-injury
* ASIA Scale A, B, or C injury at or above neurological level T4
* able to follow directions
* wheelchair users
* leg muscles responsive to stimulation

Exclusion Criteria:

* BP >140/90 mmHg to exclude for hypertension (though rare in those with high level SCI)
* current tobacco users
* significant arrhythmias
* coronary disease
* diabetes
* renal disease
* cancer
* epilepsy
* current use of cardioactive medications (except medication to support blood pressure)
* current grade 2 or greater pressure ulcers at relevant contact sites
* other neurological disease
* peripheral nerve compressions or rotator cuff tears that limit the ability to row
* history of bleeding disorders
* current use of buspirone
* pregnancy
* contraindications to Buspirone (taking MAO inhibitors, known hypersensitivity to buspirone, benzodiazepine dependence, akathisia, renal impairment, hepatic disease)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in baseline aerobic exercise capacity | Baseline, 3 months, 6 months
  Participants perform incremental FES rowing exercise test to determine maximum oxygen consumption (VO2 peak)
Change in baseline ventilation during exercise | Baseline, 3 months, 6 months
  Participants perform incremental FES rowing exercise test to determine ventilation during exercise (VE peak).

SECONDARY OUTCOMES:
Change from baseline in glucoregulatory status | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure the homeostasis model assessment (HOMA) of insulin resistance.
Change from baseline in glucoregulatory status | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure the quantitative insulin check index (QUICKI).
Change from baseline in glucoregulatory status | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure hemoglobin A1c.
Change from baseline in serum lipids | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure plasma total cholesterol.
Change from baseline in serum lipids | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure low-density lipoprotein cholesterol.
Change from baseline in serum lipids | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure high density apolipoprotein cholesterol.
Change from baseline in serum lipids | Baseline, 3 months, 6 months
  Blood will be taken via standard venipuncture to measure triglycerides.
Change from baseline in visceral adiposity | Baseline, 3 months, 6 months
  The investigators will use a 5th generation General Electric Healthcare dual x-ray absorptiometry (DXA) scanner for regional fat measurements, the DXA software can be used to define standard regions that will allow comparability of measurements throughout the study.
Change in baseline forced vital capacity | Baseline, 3 months, 6 months
  Spirometry will be used to measure lung function, specifically forced vital capacity (FVC).
Change in baseline maximal voluntary ventilation | Baseline, 3 months, 6 months
  Spirometry will be used to measure lung function, specifically maximal voluntary ventilation (MVV).
Change in baseline forced expiratory capacity in the first second | Baseline, 3 months, 6 months
  Spirometry will be used to measure lung function, specifically forced expiratory capacity in the first second (FEV1).

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States